CLINICAL TRIAL: NCT00752739
Title: Phase II Chemoprevention Trial of Selenium and Prostate Cancer (Watchful Waiting With Selenium Trial)
Brief Title: Selenium in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 97-0395-01; R01CA079080 (NIH); P30CA023074 (NIH); UARIZ-97-0395; UARIZ-HSC-97-57; DAMD17-98-1-8580; 97-0395-01
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenium

ARMS (3):
- Arm I (Placebo Comparator): Patients receive oral placebo once daily for 48 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo
- Arm II (Experimental): Patients receive low-dose oral selenium once daily for 48 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: selenium
- Arm III (Experimental): Patients receive high-dose oral selenium once daily for 48 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: selenium

INTERVENTIONS:
Dietary Supplement: selenium — Given orally
  Arms: Arm II; Arm III
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Selenium may prevent or slow the growth of prostate cancer.

PURPOSE: This randomized phase II trial is studying how well selenium works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the ability of selenium to prevent progression in patients with adenocarcinoma of the prostate.
* To investigate the ability of selenium to effectively modulate biomarkers of prostate cancer.
* To determine if selenium modifies the progression of prostate cancer based on an analysis of initial biopsy, subsequent blood biomarkers, and urological symptoms.
* To further establish the safety of chronic supplementation with selenium in these patients.

OUTLINE: Patients are stratified according to Gleason score (low vs moderate). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral placebo once daily for 48 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive low-dose oral selenium once daily for 48 months in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive high-dose oral selenium once daily for 48 months in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected periodically for biomarker laboratory studies. Blood samples are analyzed for levels of prostate-specific antigen, chromogranin A, alkaline phosphatase, alpha tocopherol, lycopene, and other vitamins; levels of selenium by atomic absorption spectrometry; and oxidative damage to DNA. Tissue samples are analyzed for levels of Bcl-2, p53, Ki-67, thioredoxin reductase, thioredoxin, and glutathione peroxidase by immunohistochemistry and for apoptotic index by TUNEL assay.

Patients complete urological symptom questionnaires and other questionnaires periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven adenocarcinoma of the prostate within the past 48 months
* Prostate-specific antigen < 50 ng/mL
* Gleason score < 8
* Currently undergoing "watchful waiting" for prostate cancer
* No metastatic disease

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 years
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 1.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No other malignancy within the past 5 years, except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

* No prior hormone therapy, radiotherapy, chemotherapy, or surgery for prostate cancer
* At least 90 days since prior and no concurrent selenium (as a dietary supplement or as part of a multivitamin) exceeding 50 mcg/day

Max Age: 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2002-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Rate of rise in serum prostate-specific antigen
Rate of rise in chromogranin A and alkaline phosphatase
Disease progression

SECONDARY OUTCOMES:
Time to prostate cancer therapy
Time to metastases
Symptoms of selenium toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R. Ahmann, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States